CLINICAL TRIAL: NCT03117777
Title: Group Cognitive Behavioral Therapy for Insomnia (CBT-I) in OIder Adults: the Clinical Outcomes of a Pilot Project
Brief Title: Group Cognitive Behavioral Therapy for Insomnia in Older Adults
Status: Withdrawn | Type: Observational
Why Stopped: REB approval denied
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Other Study IDs: 3763
Record Dates: First submitted 2017-04-10; First posted 2017-04-18 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: group cognitive behavioral therapy for insomnia — cognitive behavioral therapy for insomnia delivered in group setting for older adults

SUMMARY:
This is a quality assurance project to evaluate a therapy program offered to patients in Sleep Disorders Clinic. Group Cognitive Behavioral Therapy for Insomnia (CBT-I) is being offered to older adults. The study will consist of analyzing outcomes of a clinical program. As part of standard clinical process, patients complete measurements of sleep, daytime functioning, fatigue, quality of life, depression and anxiety symptoms before and after the treatment. The proposed study will pool and quantitatively analyze the existing clinical data. Only those program participants who consent to have their data pooled in the data analysis will be considered research subjects. Those patients who decline to have their individual data included in the analysis will continue in the therapeutic group as per usual clinical care standards.

CBT-I is a gold standard treatment for people suffering from insomnia but it is difficult to access due to a shortage of trained therapists. Insomnia prevalence increases with age and is a common sleep disturbance in the elderly. Offering the group treatment can increase access and reduce healthcare costs associated with sleep problems in the elderly.

DETAILED DESCRIPTION:
Insomnia is a sleep disorder defined as difficulty initiating or maintaining sleep at least 3 nights per week for at least 3 months and is associated with daytime impairment. The prevalence of insomnia is high, approximately 10% in the general population. Symptoms of insomnia (i.e. sleep difficulties in the absence of a full diagnosis) are even more common, with prevalence higher than 30%. The rate of insomnia symptoms in elderly populations is even higher, with approximately 50% of older adults regularly complaining about significant sleep disturbances.

Over the age of 50 years, the likelihood of a sleep problem increases as a result of a number of factors. Changes to the circadian rhythm can lead to falling asleep and waking earlier than desired. Deep sleep decreases with age, as a result nightly awakenings become more common. Co-morbidities causing nocturnal urination and joint pain can also affect sleep in older adults. These common sleep changes, along with environmental and psychological factors, can precipitate insomnia. Once disturbed sleep occurs, cognitive and behavioral factors such as dysfunctional beliefs about sleep or maladaptive sleep habits can perpetuate insomnia.

Sleep disturbance in older adulthood is associated with negative consequences across broad areas of functioning. For example, cognitive problems resulting from sleep disturbance can include increased difficulty with attention, memory and response time. Physical issues such as increased pain, falls and increased mortality rates are also associated with sleep disturbance in the elderly.

Due to the sizeable increase in sleep disturbances and the associates risks in older adults, access to safe and effective treatment becomes imperative. The increasing numbers of older adults in the general population ("the rising tide") will create a demand for practical means of delivering the necessary healthcare in a sustainable and practical way.

Medication (i.e. sedative hypnotics) may improve sleep parameters in elderly populations, however sleep problems generally resurface after discontinuation of medication. Additionally, the risk of adverse events created by sedative hypnotics, such as gait disturbance and cognitive impairment, is significant. Primarily due to the high risks associated with sedative hypnotics, they are not recommended as a fist-line treatment for insomnia. In situations where sedative hypnotics are prescribed, the recommended use duration is maximum 2 weeks.

The recommended treatment for insomnia, endorsed by clinical guidelines (e.g. the Canadian Medical Association and the American Academy of Sleep Medicine) is Cognitive Behavioural Therapy for Insomnia (CBT-I). CBT-I is also endorsed as a first-line treatment for seniors. CBT-I programs for seniors have been found to be effective in significantly increasing both sleep quality and sleep quantity.

Despite their effectiveness, CBT-I programs are often inaccessible due to Canada-wide limited resources and lack of trained professionals. CBT-I group programs have been introduced as a strategy for increasing access to insomnia treatment. Group programs fr the general adult population have been found to be similarly effective when compared with individual CBT-I, supporting this format for treatment.

Older adults have been shown to have unique sleep problems and sleep needs, and there is evidence of a good treatment response in individual therapy, however the effectiveness of group CBT-I has not been evaluated with this population. With the increased prevalence of insomnia in older adults, it is important that safe and effective treatment be available. The proposed project will therefore involve pilot testing of a group CBT-I program for seniors. It is hypothesized that seniors will improve in subjective sleep quality and sleep quantity after completing the intervention.

Research Question:

Is group CBT-I acceptable as a treatment of late-life insomnia, and does it result in subjective sleep improvements?

Methods:

The group therapy will take place in Sleep Disorders Clinic and will be offered to patients with insomnia referred from the community. The CBT-I groups will contain 6-10 patients each and will be run 10 times over a period of 24 months, for a maximum of 60 patients.

This is a quality assurance project to evaluate a therapy program offered to patients in Sleep Disorders Clinic. Group Cognitive Behavioral Therapy for Insomnia (CBT-I) is being offered to older adults. The study will consist of analyzing outcomes of a clinical program. As part of standard clinical process, patients complete measurements of sleep, daytime functioning, fatigue, quality of life, depression and anxiety symptoms before and after the treatment. The proposed study will pool and quantitatively analyze the existing clinical data. Only those program participants who consent to have their data pooled in the data analysis will be considered research subjects. Those patients who decline to have their individual data included in the analysis will continue in the therapeutic group as per usual clinical care standards.

ELIGIBILITY:
Inclusion Criteria:

* patients 65 years and older meeting diagnostic criteria for insomnia

Exclusion Criteria:

* significant physical or cognitive impairment that prevent the patients from participating in behavioural intervention (e.g. getting out of bed on their own) or cognitive intervention (e.g. learning sleep psychoeducation)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients 65 years of age and older, who meet diagnostic criteria for insomnia disorder defined as difficulty initiating or maintaining sleep associated with daytime impairment, occurring at least 3 nights per week for at least 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-10 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index | 5 months
  a validated questionnaire to assess severity of insomnia symptoms, 7 items
Pittsburgh Sleep Quality Index | 5 months
  a validated questionnaire about quality of sleep, 19 items
Epworth Sleepiness Scale | 5 months
  a validated questionnaire about level of daytime sleepiness, 8 items
Dysfunctional Beliefs and Attitudes about Sleep Questionnaire | 5 months
  a validated questionnaire to assess the patients core beliefs about their sleep, 16 items
Sleep logs | 5 months
  standard instrument used in cognitive behavioral therapy of insomnia, patient fills out data regarding sleep duration and time-in-bed duration, time to sleep onset, time awake after sleep onset, allows to evaluate sleep patterns and calculate sleep efficiency

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | 5 months
  14 item scale to assess feelings of anxiety and depression
Short Forms Health Survey SF-36 | 5 months
  quality of life measure
patient satisfaction survey | 5 months
  investigator developed brief questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata rajda, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Sleep Disorders Clinic and Laboratory, QEII Health Sciences Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No